CLINICAL TRIAL: NCT02230072
Title: Minimally Invasive Fetal Neural Tube Defect Repair Study
Brief Title: Fetoscopic Meningomyelocele Repair Study
Acronym: fMMC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael A Belfort, Professor and Chairman, Department of Obstetrics and Gynecology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-34680
Record Dates: First submitted 2014-08-22; First posted 2014-09-03 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Neural Tube Defect
Keywords: myelomeningocele; MMC; NTD; neural; defect; Spina bifida; Neural Tube Defect
MeSH Terms: conditions — Neural Tube Defects; Meningomyelocele; Spinal Dysraphism | interventions — Fetoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- fetoscopic surgical repair (Experimental): Single arm study. All patients will receive the fetoscopic repair.
  Interventions: Device: fetoscopy

INTERVENTIONS:
Device: fetoscopy — The fetoscopic arm is described above. All patients will have a laparotomy, exteriorization of the uterus, and a fetoscopic repair of the fetal open neural tube defect.
  Other Names: Karl Storz, Tuttlingen, Germany; Richard Wolf Medical Instruments, Corp.; Karl Storz Endoscopy-America, Inc.; Cook Medical, Inc.; Lexion Medical, LLC.; Terumo Pinnacle

SUMMARY:
The purpose of the study is to evaluate the maternal and fetal outcomes of a new technique for the fetoscopic repair of fetal MMC at Texas Children's Hospital Pavilion for Women.

The investigators hypothesis is that this minimally invasive technique is feasible, and that this approach will have the same efficacy as open fetal surgery for MMC, but with significantly less maternal-fetal risk. Both mother and baby will benefit from the surgery. The fetus will have a repaired MMC defect, and the mother will not have a uterine incision (hysterotomy). A hysterotomy increases the risk of uterine rupture and requires that all subsequent deliveries are by cesarean section. There may also be a decreased risk of Pre-term Premature Rupture Of Membranes (PPROM) and prematurity when compared with the current open operation. Finally, a vaginal delivery is possible following the fetoscopic fetal surgery if the baby is shown to have a skin covered repair.

DETAILED DESCRIPTION:
Spina bifida can be a devastating neurological congenital anomaly . It results from incomplete closure of the neural tube between 22 and 28 embryological days. Its incidence is approximately 1-2 per 1,000 births. It is considered the most common congenital anomaly of the central nervous system that is compatible with life.

1. The most frequent form is myelomeningocele (MMC), characterized by the extrusion of the spinal cord into a sac filled with cerebrospinal fluid (CSF), and is associated with lower limb paralysis and bowel and bladder dysfunction.
2. The majority of MMCs can be diagnosed between 14 and 20 weeks of gestation. MMC is associated with Chiari II malformation, which includes a constellation of anomalies such as hindbrain herniation, brainstem abnormalities, low-lying venous sinuses and a small posterior fossa.The Chiari II malformation can have deleterious effects on motor, cranial nerve and cognitive functions. Postnatally most MMC patients develop hydrocephalus and require a ventriculoperitoneal shunt. Shunts require lifelong monitoring and have a high failure rate due to infection, obstruction, and fracture.

Experimental studies using animal models have shown that prenatal coverage of a spina bifida-like lesion can preserve neurological function and reduce or reverse hindbrain herniation.These studies suggest a "two-hit" hypothesis in which the ultimate neurologic deficit results from a combination of the failure of normal neural-tube closure (first hit) with secondary spinal cord injury resulting from prolonged exposure of sensitive neural elements to the amniotic fluid (second hit mechanism).

Based on this hypothesis, open fetal surgical repair of MMC was proposed, and the recent publication of the NICHD sponsored randomized controlled trial demonstrated clear neonatal benefit of open in-utero fetal surgical repair of MMC. The study showed a reduction in the incidence of hydrocephalus and in the radiographic severity of hindbrain herniation (relative risk: 0.67; 95% confidence interval: 0.56-0.81).

Open in-utero fetal surgery is not without risk and the NICHD study (MOMS Trial) showed an elevation in maternal-fetal morbidity/risk when compared to the postnatally treated group, including higher risk for chorioamniotic separation (26% vs. 0%, respectively), maternal pulmonary edema (6% vs. 0%), oligohydramnios (21% vs. 0%), placental abruption (6% vs. 0%), spontaneous membrane rupture (46%; RR: 6.15; 95% CI: 2.75-13.78), spontaneous labor (38%; RR: 2.80, 95%CI: 1.51-5.18), maternal blood transfusion (9%; RR: 7.18; 95%CI: 0.90-57.01), and preterm delivery before 34 weeks (46%; RR: 9.2; 95%CI: 3.81-22.19). The reason for the increased incidence of these complications is related to the nature of the open fetal procedure, which involves a multi-faceted invasive approach including maternal laparotomy, large hysterotomy with uterine edge stapling, and open fetal repair of the spina bifida defect that may involve manipulation and exposure of the fetus for a significant amount of time.

Fetal endoscopic surgery has progressed rapidly over the past decades and the investigators are now able to perform a number of intricate procedures inside the uterus with specially designed instruments. These procedures include laser therapy for Twin-twin-transfusion syndrome, fetal cystoscopy and fulguration of posterior urethral valves, release of amniotic bands, and placement of various shunts and balloons inside fetal structures and cavities (peritoneal, pleural, cardiac, and trachea).

Fetoscopy offers a less invasive therapeutic option that could reduce a number of the morbidities (both maternal and fetal) related to open fetal procedures.

A few animal studies and some clinical human experience with fetoscopic repair of MMC have been reported showing the feasibility of covering the defect with a patch and sealant, or even in performing a full repair. These repairs have been accomplished using at least two (and sometimes more) entry ports through the uterine wall. Kohl et al. in Germany, have demonstrated the feasibility of performing a complete percutaneous fetoscopic repair of MMC using carbon dioxide to distend the uterus and provide a dry working area for the surgeon to perform the repair.

These investigators described a two-layer covering technique using an absorbable patch (Durasis, Cook, Germany) and sutures. However, while they showed that the procedure is feasible, their percutaneous technique with complete two layer surgical closure of the defect using sutures was associated with prolonged operative time and significant maternal and obstetrical morbidities.

Fetoscopy in a CO2 gas filled uterus has been recently reported by groups in Bonn, Germany (Kohl et al) and Sao Paulo, Brazil (Pedreira et al). The fetoscopic technique the investigators use has been developed and tested in a fetal sheep model of MMC by the investigators group and others (Peiro et al).

This fetoscopy technique has evolved over time to a 2-port technique developed by our team in Houston, Texas and its feasibility and applicability to the human uterus and fetus have been demonstrated and published (Belfort et al, 2017) and demonstrate an improved degree of flexibility in terms of access to the fetus regardless of placental location. The technique is designed to decrease the maternal risks of open uterus fetal surgery while maintaining a similar level of fetal benefit as seen in the MOMS trial.

The investigators technique employs an open abdomen/exteriorized (but closed) uterus methodology that allows the minimally invasive multi-layer closure of the fetal neural tube using the same closed skin repair currently employed at Baylor College of Medicine/Texas Children's Fetal Center using the open uterus approach. The technique employs a novel approach to low pressure uterine distention using the same carbon dioxide gas 8-12 mmHg that others attempting fetoscopic repair have used, but employing a much lower gas flow rate and pressure. In addition, our technique (as compared with the percutaneous method) allows improved access to the fetus in anterior placentation, ability to manipulate and maintain the fetus in the required position, and optimal port placement resulting from the exteriorized maternal uterus.

In addition, because of the exteriorized uterus and the optimal placement this allows, we require only two access ports and these can be sutured into the uterus allowing a closed seal and minimizing gas leakage. The use of humidified, warmed CO2, which we pioneered in fetal surgery, decreases membrane disruption and may prolong gestation without rupture of the membranes. Finally, recent advances in miniature surgical instruments (Storz 1.5 - 3mm surgical sets) allow unprecedented flexibility which enables a full surgical repair to be performed via a fetoscopic approach.

In preparation for the human trial we were able to perform, in a sheep model, dual access port fetoscopic neural tube closure using a 12 F cannula, a second 9F cannula, a cover patch, and a medical sealant with similar results to that seen with open fetal surgical repair in the same sheep model.26

We have now completed almost 50 cases using our 2 port exteriorized technique with results that are reflect our initial hypothesis (Belfort et al , 2017). As with any technique there have been advances in instrumentation and technique and the study is ongoing investigating the multilayer closure technique.

In this protocol, the repair of the open neural tube defect will follow the same principles as we use in open repairs currently being done at this institution. This involves release of the placode, dissection of the surrounding skin and attempted primary closure of the defect using a Durepair patch, a muscle or duro-fascial flap, and available skin. In those cases where we are able to complete the procedure with full skin closure of the defect, the only difference between the open uterus procedure and the fetoscopic procedure, will be that the surgery will be done fetoscopically rather than through an open uterine incision. If we are unable to close the skin primarily despite best fetoscopic efforts, the option of performing/completing the repair as an open procedure exists and will be offered to the patient. The patient is monitored in hospital until ready for discharge.

Approximately 6 weeks after the surgery a post-procedure fetal MRI will be performed. If there is evidence of good closure of the neural tube defect and reversal of the Chiari II malformation, a vaginal delivery can be attempted based on obstetric criteria. Patients will be followed in person every 3-4 months after birth to 12 months at the Spina Bifida Clinic at TCH. Remaining visits will be yearly up to 5 years. If this is not possible, questionnaire(s) will be mailed to the child's parents and records will be requested from the treating neurosurgeon on this same schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women - maternal age 18 years or older and capable of consenting for their own participation in this study,
2. Singleton pregnancy,
3. MMC with the upper boundary located between T1 and S1,
4. Evidence of hindbrain herniation (confirmed on MRI to have an Arnold-Chiari type II malformation),
5. Absence of chromosomal abnormalities and associated anomalies,
6. Gestational age at the time of the procedure will be between 19 0/7 weeks and 25 6/7 weeks,
7. Normal karyotype and/or normal chromosomal microarray (CMA) by invasive testing (amniocentesis or CVS). If there is a balanced translocation with normal MCA with no other anomalies the candidate can be included. Patients declining invasive testing will be excluded.
8. Family has considered and declined the option of termination of the pregnancy at less than 24 weeks,
9. Family meets psychosocial criteria (sufficient social support, ability to understand requirements of the study), and
10. Parental/guardian permission (informed consent) for follow up of child after birth.

Exclusion Criteria:

1. Fetal anomaly unrelated to MMC,
2. Severe kyphosis,
3. Increased risk for preterm labor including short cervical length (<1.5 cm), history of incompetent cervix with or without cerclage, and previous preterm birth,
4. Placental abnormalities (previa, abruption, accreta) known at time of enrollment,
5. A pre-pregnancy body-mass index ≥40,
6. Contraindications to surgery including previous hysterotomy (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, major myomectomy resection, or previous fetal surgery) in active uterine segment,
7. Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, and uterine anomalies,
8. Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy,
9. Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment,
10. Maternal medical condition that is a contraindication to surgery or anesthesia,
11. Low amniotic fluid volume (Amniotic Fluid Index less than 6cm) if deemed to be due to fetal anomaly, poor placental perfusion or function, or membrane rupture. Low amniotic fluid volume that responds to maternal hydration is not an exclusion criterion,
12. Patient does not have a support person (e.g. Spouse, partner, mother) available to support the patient for the duration of the pregnancy,
13. Inability to comply with the travel and follow-up requirements of the trial,
14. Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy, and
15. Patient scores as severely depressed on the BDI-II questionnaire; a score of 29 or above.
16. Maternal hypersensitivity to collagen.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Feasibility | Time of procedure
  Whether the minimally invasive technique can be technically performed in human patients (success of primary skin closure) in a safe and effective manner.

SECONDARY OUTCOMES:
Reversal of the Chiari II malformation with complete closure of the spinal defect. | at birth
  Whether the minimally invasive technique results in an acceptable fetal outcome as defined by reversal of the Chiari II malformation, a reduced need for ventriculoperitoneal shunting or other procedures to avoid or treat hydrocephalus, and complete closure of the spinal defect with protection of the placode. In addition the procedure will be assessed as to whether it prevents loss of neurological level during intra-uterine life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Belfort, M.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Stanford University: Lucille Packard's Childrens Hospital, Stanford, California
  - Texas Childrens Hospital, Houston, Texas

REFERENCES:
- [Derived] Corroenne R, Mehollin-Ray AR, Johnson RM, Whitehead WE, Espinoza J, Castillo J, Castillo H, Orman G, Donepudi R, Huisman TAGM, Nassr AA, Belfort MA, Sanz Cortes M, Shamshirsaz AA. Impact of the volume of the myelomeningocele sac on imaging, prenatal neurosurgery and motor outcomes: a retrospective cohort study. Sci Rep. 2021 Jun 23;11(1):13189. doi: 10.1038/s41598-021-92739-2. PMID 34162982
- [Derived] Belfort MA, Whitehead WE, Shamshirsaz AA, Bateni ZH, Olutoye OO, Olutoye OA, Mann DG, Espinoza J, Williams E, Lee TC, Keswani SG, Ayres N, Cassady CI, Mehollin-Ray AR, Sanz Cortes M, Carreras E, Peiro JL, Ruano R, Cass DL. Fetoscopic Open Neural Tube Defect Repair: Development and Refinement of a Two-Port, Carbon Dioxide Insufflation Technique. Obstet Gynecol. 2017 Apr;129(4):734-743. doi: 10.1097/AOG.0000000000001941. PMID 28277363